CLINICAL TRIAL: NCT06173921
Title: Comparing Accuracy of Static Navigation Systems and Robotic System in Partially Edentulous in Posterior Area: A Randomized Clinical Trial
Brief Title: The Accuracy of Static Navigation Systems and Robotic System in Partially Edentulous in Posterior Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Ke Song, Principal Investigator, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ-IRB20231192
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Dental Implant
Keywords: Dental implant; Robotic system; Static navigation system

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic system (Experimental): implant placement by robotic surgery
  Interventions: Procedure: robotic system
- Static system (Active Comparator): implant placement by static navigation surgery
  Interventions: Procedure: Static navigation system

INTERVENTIONS:
Procedure: robotic system — Implant placement will be navigated by robotic system based on a digital plan
  Arms: Robotic system
Procedure: Static navigation system — Implant placement will be navigated by static navigation system based on a digital plan
  Arms: Static system

SUMMARY:
The aim of this randomized clinical trial to compare the implant positional accuracy of robotic system-assisted implant surgery with that of static system-assisted implant surgery. Patients will be recruited and randomly assigned to either the robotic surgery group or the static navigation surgery group to evaluate the accuracy of the implants in both groups and to compare patient-reported and physician-reported outcomes of the two approaches.

DETAILED DESCRIPTION:
Dental implants have been widely used for replacing the lost natural teeth, with evidence of long-term success and improvement of patients' quality of life. Nevertheless, proper implant position is considered today an essential prerequisite for ensuring successful treatment outcomes, as well as long-term maintenance of the prosthesis and the peri-implant tissue health.Therefore, we plan to conduct this randomized clinical trialto compare the implant positional accuracy of robotic system-assisted implant surgery with that of static system-assisted implant surgery. Patients will be recruited and randomly assigned to either the robotic surgery group or the static navigation surgery group to evaluate the accuracy of the implants in both groups and to compare patient-reported and physician-reported outcomes of the two approaches.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed voluntarily.
* Aged at least 18 years.
* Partial edentulousness in the posterior maxillary or mandibular region (premolar, molar, maximum two in a row).
* Sufficient bone volume for implant placement without bone augmentation;
* The minimum number of residual teeth was seven teeth.
* Good communication with the physician, compliance, ability to follow the physician's advice to maintain oral hygiene.

Exclusion criteria:

* Systemic disease that would interfere with dental implant surgery.
* Bisphosphonate treatment.
* Untreated, uncontrolled periodontal disease.
* Heavy smoker (more than 10 cigarettes per day).
* Poor oral hygiene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
implant positional accuracy | immediately after surgery
  The implant placement accuracy was measured by overlapping the planned position of the implant in the preoperative CBCT and its final position assessed through a postoperative CBCT.

SECONDARY OUTCOMES:
Pain perception | immediately after surgery, and 1 to 7 days after surgery.
  patient pain perception after surgery will recorded by visual analogue scale (VAS with range from 0 to 10 with 10 being the highest possible pain experience)
Surgery complication | Immediately and 7 days after surgery
  Complication related to implant placement surgery.

IPD SHARING:
Plan to Share IPD: No